CLINICAL TRIAL: NCT03780283
Title: Efficacy and Safety of Anlotinib as Maintenance Treatment After First-line Chemotherapy in Small Cell Lung Cancer（SCLC）：a Phase II Study
Brief Title: Efficacy and Safety of Anlotinib as Maintenance Treatment After First-line Chemotherapy in SCLC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: First Hospital of Shijiazhuang City (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LC02
Record Dates: First submitted 2018-12-17; First posted 2018-12-19 (Actual); Last update posted 2018-12-21 (Actual); Status verified 2018-12

CONDITIONS: Carcinoma; Lung Neoplasm; Small Cell Lung Cancer
Keywords: SCLC; maintenance; Anlotinib
MeSH Terms: conditions — Carcinoma; Lung Neoplasms; Small Cell Lung Carcinoma | interventions — anlotinib

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anlotinib Hydrochloride (Experimental): Participants receive Anlotinib 12mg, administered as PO on Day1-14 of each 21-day cycle until documented PD
  Interventions: Drug: Anlotinib Hydrochloride
- placebo (No Intervention): observation

INTERVENTIONS:
Drug: Anlotinib Hydrochloride — Participants receive Anlotinib 12mg, administered as PO on Day1-14 of each 21-day cycle until documented PD or had unacceptable toxicity
  Other Names: Anlotinib
  Arms: Anlotinib Hydrochloride

SUMMARY:
Investigations prospectively collected the SCLC patients who received current standard first-line treatment, the response was not progression disease(PD). and then participants receive Anlotinib 12mg, administered as PO on Day1-14 of each 21-day cycle until documented PD or had unacceptable toxicity. This regimen is compared to the effects a observation without treatment after the first-line therapy. The aim of the study is therefore to evaluate the efficacy and safety of Anlotinib as maintenance treatment after first-line chemotherapy in SCLC patients.

ELIGIBILITY:
Inclusion Criteria:

* 1. The subjects volunteered to participate in this study and signed the informed consent form, with good compliance and follow-up.

  2. Male or female patients aged 18-75 years old. 3.After receiving the current standard first-line treatment, patients with small-cell Lung cancer who have received non-surgical treatment have reached stable disease(SD), (partial remission)PR and (complete remission)CR patients (a limit or extensive stage according to Veterans Administration Lung Study Group (VALG)).

  4. Has a life expectancy of at least 3 months. 5. Has a performance status of 0 or 2 on the Eastern Cooperative Oncology Group (ECOG) Performance Status.

  6.Has adequate organ function. 7. Patients with asymptomatic or mild brain metastasis may be enrolled. 8. If female of childbearing potential, is willing to use adequate contraception for the course of the study through 120 days after the last dose of study medication or through 180 days after last dose of chemotherapeutic agents.

  9. If male with a female partner(s) of child-bearing potential, must agree to use adequate contraception starting with the first dose of study medication through 120 days after the last dose of study medication or through 180 days after last dose of chemotherapeutic agents.

Exclusion Criteria:

* 1.Non-small Cell Lung cancer 2. Imaging (CT or MRI) showed that the central tumor invaded the large blood vessels; or there is obvious pulmonary cavitation or necrotic tumor; 3.History and complications 3.1 Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis.(patients with brain metastasis who have completed treatment 14 days before enrollment and have stable symptoms can be included in the group, but they need to be confirmed as having no symptoms of cerebral hemorrhage by brain MRI, CT).

3.2 Have Participated in other clinical studies or less than 4 weeks before the end of treatment in the previous clinical study.

3.3 Other active malignancies requiring concurrent treatment. 3.4 Known history of prior malignancy except if participant has undergone potentially curative therapy with no evidence of that disease recurrence for 5 years since initiation of that therapy, except for successful definitive resection of basal cell carcinoma of the skin, superficial bladder cancer, squamous cell carcinoma of the skin, in situ cervical cancer, or other in situ cancers.

3.5 Patients who have not recovered to level 1 or lower of The Common Terminology Criteria for Adverse Events 4.0 （NCI-CTCAE4.0）. After previous systemic anti-tumor treatment with anti-tumor treatment-related adverse reactions (except hair loss).

3.6 Abnormal coagulation function international normalized ratio(INR) >1.5 or prothrombin time(PT) > ULN+4 s or activated partial thromboplastin time (APTT) > 1.5ULN), with bleeding tendency or receiving thrombolytic or anticoagulant treatment.

3.7 Is expected to require any other form of antineoplastic therapy while on study.

3.8 Received a live-virus vaccination within 30 days of planned start of study medication.

3.9 Known sensitivity to any component of Anlotinib. 3.10 Has active autoimmune disease that has required systemic treatment in past 2 years.

3.11 Is on chronic systemic steroids. 3.12 Has an active infection requiring therapy. 3.13 Has known history of Human Immunodeficiency Virus (HIV). 3.14 Has known active Hepatitis B or C. 3.15 Has known psychiatric or substance abuse disorder that would interfere with cooperation with the requirements of the trial.

3.16 Is a regular user (including "recreational use") of any illicit drugs or had a recent history (within the last year) of substance abuse (including alcohol).

3.17 Has symptomatic ascites or pleural effusion. 3.18 Has interstitial lung disease or a history of pneumonitis that required oral of IV glucocorticoids to assist with management.

3.19 Two or more combination therapies for hypertension that are still uncontrollable (systolic blood pressure greater than 140 mmHg or diastolic blood pressure greater than 90 mmHg).

3.20 Arteriovenous thrombosis events occurred within 12 months before enrollment, such as cerebrovascular accidents (including temporary ischemic attack, cerebral hemorrhage, cerebral infarction), deep vein thrombosis and pulmonary embolism.

3.21 Clinically significant hemoptysis occurred within 3 months before enrollment (hemoptysis > 50ml daily);Or bleeding symptoms of significant clinical significance or with a clear bleeding tendency, such as gastrointestinal bleeding, bleeding gastric ulcer, baseline stool occult blood ++ or above, or suffering from vasculitis.

3.22 Factors that significantly affect oral drug absorption, such as inability to swallow, chronic diarrhea and intestinal obstruction.

3.23 Is pregnant or breast feeding, or expecting to conceive or father children prior to 120 days after the last dose of study medication or through 180 days after last dose of chemotherapeutic agents.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2020-01-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | Up to 6 months
  PFS was defined as the time from randomization to documented disease progression per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) or death due to any cause, whichever occurred first and was based on blinded independent central radiologists' (BICR) review. Progressive Disease (PD) was defined as ≥20% increase in the sum of diameters of target lesions and an absolute increase of ≥5 mm. (Note: the appearance of one or more new lesions was also considered progression). Participants were evaluated every 9 weeks with radiographic imaging to assess their response to treatment.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | 24 months
  ORR was defined as the percentage of participants in the analysis population who experienced a Complete Response (CR; disappearance of all target lesions) or a Partial Response (PR; at least a 30% decrease in the sum of diameters of target lesions) and was assessed using RECIST 1.1 based on BICR evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Zhang, M.D., Study Chair — The First Hospital of Shijiazhuang
Locations (1):
- The First Hospital of Shijiazhuang, Shijiazhuang, Hebei, China